CLINICAL TRIAL: NCT07183839
Title: Immersive Virtual Reality Induces Procedural Analgesia, Anxiolysis and Anterograde Amnesia:A Randomized Controlled Study 2
Brief Title: The Effect of Immersive VR Distraction on Memory: Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Research Scientist at the UW Dept of Mechanical Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VRAnalgesia2025b
Record Dates: First submitted 2025-09-10; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Virtual Reality Amnesia
Keywords: immersive virtual reality distraction,; memory; see through VR

STUDY DESIGN:
Who Masked: Participant
Masking Description: The use of a plausible control condition helped mask the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Tech virtual reality (Experimental): Participants used their cyberhands to interact with virtual objects while in immersive virtual reality, while they listen to and memorize a list of 15 study words rea to them from the real world.
  Interventions: Behavioral: Immersive Virtual Reality
- Low Tech VR (Sham Comparator): Participants wore an Apple Vision Pro VR goggles that allowed them to see the real world in their VR goggles, via video streaming from cameras mounted on the VR helmet, while memorizing a list of words they heard from the real world.
  Interventions: Behavioral: Plausible control condition

INTERVENTIONS:
Behavioral: Immersive Virtual Reality — While wearing an immersive VR helmet, participants grabbed virtual objects andd put them into a bowl of virtual water, while memorizing a list of words from the real world.
  Arms: High Tech virtual reality
Behavioral: Plausible control condition — Participant passively viewed the laboratory room they saw while wearing Apple Vision Pro goggles, while memorizing a list of words read to them from the real world.
  Arms: Low Tech VR

SUMMARY:
This study measures how many words people can recall. Some words are studied/heard/learned while in immersive Virtual Reality, and some are studied/heard/learned while in a plausible control distraction.

DETAILED DESCRIPTION:
In this Study (n=20), participants recalled word lists during a plausible semi-immersive control condition (passive Apple Vision Pro see-through mode) versus during interactive immersive VR. Participants also later received brief heat pain stimuli during No VR versus immersive VR and provided pain and anxiety and distraction ratings on 0-10 graphic rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older

Exclusion Criteria:

* People who have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.
* Not enrolled in a course at the University of Washington Psychology Dept., not participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,
* Seizure history,
* Unusual sensitivity or lack of sensitivity to pain,
* Sensitive skin,
* Sensitive feet
* Migraines
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Word Recall accuracy | begin 15 seconds after the last word
  Number of study words recalled during an immediate recall task
Subjective ratings of Distraction | Measured immediately after the free recall of each word list.
  Participants rated how distracted they were in each treatment condition

SECONDARY OUTCOMES:
During Phase 2, VR pain reduction was measured | subjective pain ratings measured immediately after each brief thermal stimulus
  graphic ratings of worst pain intensity and other GRS pain ratings during brief thermal stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified summarized aggregated data will be available upon reasonable request.
Time Frame: De-identified summarized aggregated data will be available upon publication in a peer reviewed journal until 2030
Access Criteria: summarized aggregate data will be made available upon reasonable request by e-mailing the primary contact.

REFERENCES:
- [Background] Hoffman HG, Fontenot MR, Garcia-Palacios A, Greenleaf WJ, Alhalabi W, Curatolo M, Flor H. Adding tactile feedback increases avatar ownership and makes virtual reality more effective at reducing pain in a randomized crossover study. Sci Rep. 2023 May 22;13(1):7915. doi: 10.1038/s41598-023-31038-4. PMID 37217536